CLINICAL TRIAL: NCT04812938
Title: Exploiting Pathogenic Tp53 Mutation for Early Diagnosis of Ovarian Cancer by Mean of Papanicolau Test
Acronym: PAPAudit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Paolo Zola, Principal Investigator, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: PAPAudit
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; pap-test
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For each EOC patient, one FFPE biopsy from primary tumor, possibly one FFPE biopsy from a synchronous metastatic lesion will be retrieved from the Laboratory of Pathological Anatomy at each hospital center. For each FFPE sample, a minimum tumor content of 40% will be guarantee by the pathologist of the hospital who performed the diagnosis of EOC and at least three to six slides (5 micron thick) will be prepared, with the representative area of tumor marked on each slide for DNA purification. Moreover, all available patient's Pap Test smears sampled up to eight years before EOC diagnosis will be collected. All samples will be shipped to and stored at the Laboratory of Cancer Pharmacology, IRCCS Humanitas Research Hospital at under the responsibility of Dr. Sergio Marchini.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with Ovarian cancer and pap test available — Define the possibility to detect through the pap test the presence of ovarian cancer cells in vaginal smear in patients with no evidence of ginecological malignancies.

SUMMARY:
The aim of the project is to corroborate them on a large retrospective cohort of HGS-EOC and confirm the possibility of identify TP53 mutations in high grade endometrioid tumors.

This will consequently allow to confirm the previous results and define with a greater precision the temporal windows in which it will be possible to detect, through the TP53 analysis, tumor material by vaginal swab sampling. The results of the study will be the first step of a multiphase prospective validation program for the development of a novel approach for early diagnosis of EOC.

DETAILED DESCRIPTION:
All participating women will be identified through the ovarian cancer audit implemented by the "Oncological Network of Piedmont and Valle d'Aosta" and the Clinical Epidemiology Unit of CPO Piemonte between 2015 and 2020. Women with EOC, and the center where they have been treated for the tumor, will be identified by linking the databases of the "Oncological Network of Piedmont and Valle d'Aosta" with those of the "Prevenzione Serena" project.

A few clinical information from EOC patients will be collected by clinical investigators at each center using an electronic case report form (e-CRF) developed at the Mario Negri Institute. These information will include age, date of diagnosis, histological subtype and grading, tumor stage according to FIGO 2014 classification2,3, previous gynecologic conditions and surgical operations, date of Pap Test collection, and Pap Test cytological reports. Participants' data will be identified by a unique patient code.

ELIGIBILITY:
Inclusion Criteria:

age ≥18 years;

* confirmed histologic diagnosis of HGS-EOC or high grade endometrioid tumor;
* presence of one FFPE primary tumor biopsy with at least 40% of tumor cells based on Hematoxylin and Eosin staining, in the archive of the Pathology Departments of the hospital centers where they have been treated;
* presence of one or more Pap Tests sampled up to eight years before EOC diagnosis during routine cervical cancer screening;
* negative history for other gynecologic malignancies;

Exclusion Criteria:

* pap test not available in patients with ovarian cancer

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will be composed of about 190 women with a diagnosis of EOC, identified through the ovarian cancer audit conducted by the "Rete Oncologica Piemonte e Valle d'Aosta" between 2015 and 2020. In order to be eligible for the study, patients should respect the following inclusion criteria:
  * age ≥18 years;
  * confirmed histologic diagnosis of HGS-EOC or high grade endometroid tumor;
  * presence of one FFPE primary tumor biopsy with at least 40% of tumor cells based on Hematoxylin and Eosin staining, in the archive of the Pathology Departments of the hospital centers where they have been treated;
  * presence of one or more Pap Tests sampled up to eight years before EOC diagnosis during routine cervical cancer screening;
  * negative history for other gynecologic malignancies;
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2021-04-12 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that clonal pathogenic TP53 variants of HGS-EOC can be detected in patient-matched PAP tests | We can estimate six month to obtain pathological sample from the different hospital involved in this protocol and in the mean time to set up the laboratory procedures in large scale.
  To validate the preliminary data obtained by Paracchini 14, which found that the clonal pathogenic TP53 variants of HGS-EOC can be detected in PAP tests of patient tratted by ovarian cancer performed more than two years before the diagnosis of ovarian neoplasia.
  Within this aim, we will calculate the detection rate and define the temporal window up to which the detection of the TP53 variant is feasible and set up the optimal experimental conditions, such as DNA quality and quantity, that will be used in the downstream steps for the assay development.
Demonstrate that clonal pathogenic TP53 variants of HGS-EOC can be detected in patient-matched PAP tests | In the following six months the data obtained are processed. The final analisys is forecast within one year.
  The second outcome is the evaluation of the percentage of pap test negative for cervical cancer and positive for genetic determination of ovarian neoplastic cells in pre clinic stage of ovarian neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zola, MD/PhD, Principal Investigator — Department of Surgical Science University of Turin
Locations (2):
- Italy (2):
  - Department of Biomedical Sciences - Humanitas University, Milan
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin

IPD SHARING:
Plan to Share IPD: Yes
This study is part of a more complex and long-lasting project aimed to develop an innovative strategy for early diagnosis of EOC. It aims to detect TP53 variants in the DNA purified from PAP tests, as an early genetic biomarker of EOC tumorigenesis.
Supporting Information: Study Protocol
Time Frame: 12-18 months
Access Criteria: Age ≥18 years;
  * confirmed histologic diagnosis of HGS-EOC or high grade endometrioid tumor;
  * presence of one FFPE primary tumor biopsy with at least 40% of tumor cells based on Hematoxylin and Eosin staining, in the archive of the Pathology Departments of the hospital centers where they have been treated;
  * presence of one or more Pap Tests sampled up to eight years before EOC diagnosis during routine cervical cancer screening;
  * negative history for other gynecologic malignancies;
  * written informed consent for the participation to the study and the molecular analysis of biological samples.

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Reid BM, Permuth JB, Sellers TA. Epidemiology of ovarian cancer: a review. Cancer Biol Med. 2017 Feb;14(1):9-32. doi: 10.20892/j.issn.2095-3941.2016.0084. PMID 28443200
- [Result] Bast RC Jr, Matulonis UA, Sood AK, Ahmed AA, Amobi AE, Balkwill FR, Wielgos-Bonvallet M, Bowtell DDL, Brenton JD, Brugge JS, Coleman RL, Draetta GF, Doberstein K, Drapkin RI, Eckert MA, Edwards RP, Elias KM, Ennis D, Futreal A, Gershenson DM, Greenberg RA, Huntsman DG, Ji JXY, Kohn EC, Iavarone C, Lengyel ER, Levine DA, Lord CJ, Lu Z, Mills GB, Modugno F, Nelson BH, Odunsi K, Pilsworth JA, Rottapel RK, Powell DJ Jr, Shen L, Shih IM, Spriggs DR, Walton J, Zhang K, Zhang R, Zou L. Critical questions in ovarian cancer research and treatment: Report of an American Association for Cancer Research Special Conference. Cancer. 2019 Jun 15;125(12):1963-1972. doi: 10.1002/cncr.32004. Epub 2019 Mar 5. PMID 30835824
- [Result] Henderson JT, Webber EM, Sawaya GF. Screening for Ovarian Cancer: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Feb 13;319(6):595-606. doi: 10.1001/jama.2017.21421. PMID 29450530
- [Result] Menon U, Gentry-Maharaj A, Hallett R, Ryan A, Burnell M, Sharma A, Lewis S, Davies S, Philpott S, Lopes A, Godfrey K, Oram D, Herod J, Williamson K, Seif MW, Scott I, Mould T, Woolas R, Murdoch J, Dobbs S, Amso NN, Leeson S, Cruickshank D, McGuire A, Campbell S, Fallowfield L, Singh N, Dawnay A, Skates SJ, Parmar M, Jacobs I. Sensitivity and specificity of multimodal and ultrasound screening for ovarian cancer, and stage distribution of detected cancers: results of the prevalence screen of the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS). Lancet Oncol. 2009 Apr;10(4):327-40. doi: 10.1016/S1470-2045(09)70026-9. Epub 2009 Mar 11. PMID 19282241
- [Result] Jacobs IJ, Menon U, Ryan A, Gentry-Maharaj A, Burnell M, Kalsi JK, Amso NN, Apostolidou S, Benjamin E, Cruickshank D, Crump DN, Davies SK, Dawnay A, Dobbs S, Fletcher G, Ford J, Godfrey K, Gunu R, Habib M, Hallett R, Herod J, Jenkins H, Karpinskyj C, Leeson S, Lewis SJ, Liston WR, Lopes A, Mould T, Murdoch J, Oram D, Rabideau DJ, Reynolds K, Scott I, Seif MW, Sharma A, Singh N, Taylor J, Warburton F, Widschwendter M, Williamson K, Woolas R, Fallowfield L, McGuire AJ, Campbell S, Parmar M, Skates SJ. Ovarian cancer screening and mortality in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2016 Mar 5;387(10022):945-956. doi: 10.1016/S0140-6736(15)01224-6. Epub 2015 Dec 17. PMID 26707054
- [Result] Ciardiello F, Arnold D, Casali PG, Cervantes A, Douillard JY, Eggermont A, Eniu A, McGregor K, Peters S, Piccart M, Popescu R, Van Cutsem E, Zielinski C, Stahel R. Delivering precision medicine in oncology today and in future-the promise and challenges of personalised cancer medicine: a position paper by the European Society for Medical Oncology (ESMO). Ann Oncol. 2014 Sep;25(9):1673-1678. doi: 10.1093/annonc/mdu217. Epub 2014 Jun 20. No abstract available. PMID 24950979
- [Result] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Result] Vang R, Levine DA, Soslow RA, Zaloudek C, Shih IeM, Kurman RJ. Molecular Alterations of TP53 are a Defining Feature of Ovarian High-Grade Serous Carcinoma: A Rereview of Cases Lacking TP53 Mutations in The Cancer Genome Atlas Ovarian Study. Int J Gynecol Pathol. 2016 Jan;35(1):48-55. doi: 10.1097/PGP.0000000000000207. PMID 26166714
- [Result] Labidi-Galy SI, Papp E, Hallberg D, Niknafs N, Adleff V, Noe M, Bhattacharya R, Novak M, Jones S, Phallen J, Hruban CA, Hirsch MS, Lin DI, Schwartz L, Maire CL, Tille JC, Bowden M, Ayhan A, Wood LD, Scharpf RB, Kurman R, Wang TL, Shih IM, Karchin R, Drapkin R, Velculescu VE. High grade serous ovarian carcinomas originate in the fallopian tube. Nat Commun. 2017 Oct 23;8(1):1093. doi: 10.1038/s41467-017-00962-1. PMID 29061967
- [Result] Ahmed AA, Etemadmoghadam D, Temple J, Lynch AG, Riad M, Sharma R, Stewart C, Fereday S, Caldas C, Defazio A, Bowtell D, Brenton JD. Driver mutations in TP53 are ubiquitous in high grade serous carcinoma of the ovary. J Pathol. 2010 May;221(1):49-56. doi: 10.1002/path.2696. PMID 20229506
- [Result] Kinde I, Bettegowda C, Wang Y, Wu J, Agrawal N, Shih IeM, Kurman R, Dao F, Levine DA, Giuntoli R, Roden R, Eshleman JR, Carvalho JP, Marie SK, Papadopoulos N, Kinzler KW, Vogelstein B, Diaz LA Jr. Evaluation of DNA from the Papanicolaou test to detect ovarian and endometrial cancers. Sci Transl Med. 2013 Jan 9;5(167):167ra4. doi: 10.1126/scitranslmed.3004952. PMID 23303603
- [Result] Wang Y, Li L, Douville C, Cohen JD, Yen TT, Kinde I, Sundfelt K, Kjaer SK, Hruban RH, Shih IM, Wang TL, Kurman RJ, Springer S, Ptak J, Popoli M, Schaefer J, Silliman N, Dobbyn L, Tanner EJ, Angarita A, Lycke M, Jochumsen K, Afsari B, Danilova L, Levine DA, Jardon K, Zeng X, Arseneau J, Fu L, Diaz LA Jr, Karchin R, Tomasetti C, Kinzler KW, Vogelstein B, Fader AN, Gilbert L, Papadopoulos N. Evaluation of liquid from the Papanicolaou test and other liquid biopsies for the detection of endometrial and ovarian cancers. Sci Transl Med. 2018 Mar 21;10(433):eaap8793. doi: 10.1126/scitranslmed.aap8793. PMID 29563323
- [Result] Paracchini L, Pesenti C, Delle Marchette M, Beltrame L, Bianchi T, Grassi T, Buda A, Landoni F, Ceppi L, Bosetti C, Paderno M, Adorni M, Vicini D, Perego P, Leone BE, D'Incalci M, Marchini S, Fruscio R. Detection of TP53 Clonal Variants in Papanicolaou Test Samples Collected up to 6 Years Prior to High-Grade Serous Epithelial Ovarian Cancer Diagnosis. JAMA Netw Open. 2020 Jul 1;3(7):e207566. doi: 10.1001/jamanetworkopen.2020.7566. PMID 32609349
- [Result] Cybulska P, Paula ADC, Tseng J, Leitao MM Jr, Bashashati A, Huntsman DG, Nazeran TM, Aghajanian C, Abu-Rustum NR, DeLair DF, Shah SP, Weigelt B. Molecular profiling and molecular classification of endometrioid ovarian carcinomas. Gynecol Oncol. 2019 Sep;154(3):516-523. doi: 10.1016/j.ygyno.2019.07.012. Epub 2019 Jul 21. PMID 31340883
- [Result] Li H, Durbin R. Fast and accurate long-read alignment with Burrows-Wheeler transform. Bioinformatics. 2010 Mar 1;26(5):589-95. doi: 10.1093/bioinformatics/btp698. Epub 2010 Jan 15. PMID 20080505
- [Result] Cibulskis K, Lawrence MS, Carter SL, Sivachenko A, Jaffe D, Sougnez C, Gabriel S, Meyerson M, Lander ES, Getz G. Sensitive detection of somatic point mutations in impure and heterogeneous cancer samples. Nat Biotechnol. 2013 Mar;31(3):213-9. doi: 10.1038/nbt.2514. Epub 2013 Feb 10. PMID 23396013
- [Result] McLaren W, Gil L, Hunt SE, Riat HS, Ritchie GR, Thormann A, Flicek P, Cunningham F. The Ensembl Variant Effect Predictor. Genome Biol. 2016 Jun 6;17(1):122. doi: 10.1186/s13059-016-0974-4. PMID 27268795